CLINICAL TRIAL: NCT02958592
Title: Assessment of Hepatic Fibrosis by Shear Wave Elastography in Patients With Liver Malignancy: A Prospective Single-center Study
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Doctor, Sun Yat-sen University
Other Study IDs: 2016-FXY-132
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Liver Tumor; Hepatic Fibrosis
Keywords: shear-wave elastography; hepatic fibrosis; liver tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: patients with liver tumor intend to perform hepatectomy
  Interventions: Other: two-dimensional shear-wave elastography (SWE)

INTERVENTIONS:
Other: two-dimensional shear-wave elastography (SWE) — performa two-dimensional shear-wave elastography (SWE) for staging hepatic fibrosis in the background liver parenchyma in patients with liver tumors before hepatic resection

SUMMARY:
To evaluate the diagnostic performance of two-dimensional shear-wave elastography (SWE) for staging hepatic fibrosis in the background liver parenchyma in patients with liver tumors before hepatic resection, using resected tissue pathology as a reference standard.

ELIGIBILITY:
Inclusion Criteria:

* (i) patients with a solid focal liver lesion that was pathologically proven or diagnosed by imaging methods such as conventional US, CT or MR imaging; (ii) patients scheduled to undergo a hepatectomy; (iii) patients with a lesion ≥1.0 cm in diameter.

Exclusion Criteria:

* (i) patients with a history of chemotherapy; (ii) patients unable to properly hold their breath.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with liver tumor intend to hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Stage of hepatic fibrosis | within the first 7 days after surgery
  compare the stage of hepatic fibrosis between SWE test with specimens after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Minshan Chen, Study Director — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Zheng W, Zhang YJ, Xu L, Chen JB, Chen JC, Chen MS, Zhou Z. Assessing Hepatic Fibrosis Using 2-D Shear Wave Elastography in Patients with Liver Tumors: A Prospective Single-Center Study. Ultrasound Med Biol. 2017 Nov;43(11):2522-2529. doi: 10.1016/j.ultrasmedbio.2017.07.003. Epub 2017 Aug 12. PMID 28807448